CLINICAL TRIAL: NCT05009901
Title: A Pilot Study of Antioxidant Therapy (Alpha Lipoic Acid, ALA) in OSA Patients
Brief Title: A Pilot Study of Antioxidant Therapy in Obstructive Sleep Apnea Patients
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Rachel Jen, Clinical Assistant Professor, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: H20-03562
Record Dates: First submitted 2021-08-10; First posted 2021-08-18 (Actual); Last update posted 2022-05-25 (Actual); Status verified 2022-05

CONDITIONS: Obstructive Sleep Apnea of Adult
Keywords: Obstructive Sleep Apnea; Antioxidant; Alpha Lipoic Acid; Inflammation; Endothelial Function
MeSH Terms: conditions — Sleep Apnea, Obstructive; Inflammation | interventions — Thioctic Acid; Tablets

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Alpha Lipoic Acid (Experimental): alpha lipoic acid PO 600 mg daily for 8 weeks
  Interventions: Drug: Alpha Lipoic Acid 600 MG Oral Tablet
- Placebo (Placebo Comparator): placebo PO daily for 8 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Alpha Lipoic Acid 600 MG Oral Tablet — Alpha lipoic acid 600 mg daily for 8 weeks
  Other Names: Alpha lipoic acid
  Arms: Alpha Lipoic Acid
Drug: Placebo — Placebo one tablet daily for 8 weeks
  Arms: Placebo

SUMMARY:
Sleep apnea is a common under-diagnosed medical disorder, and moderate to severe disease is found in approximately 9% of men and 4% of women. The disease is characterized by repetitive collapse of the airway during sleep, causing sleep disruption, episodic low oxygen levels, and daytime sleepiness. Also, patients with sleep apnea are at high risk of developing cardiovascular disease (including strokes and heart attacks). Partly, this is because the episodic low oxygen levels followed by higher oxygen levels due to sleep apnea results in the generation of reactive oxygen species (unstable and potentially toxic substances caused by interactions with oxygen) and a state of "oxidative stress." Oxidative stress is an important contributing factor to heart disease. We are interested in determining whether treatment with antioxidants, which are substances that help reduce oxidative stress, helps cardiovascular health in patients with sleep apnea. Specifically, we want to determine whether treatment improves blood vessel function (an early sign of heart disease), and blood/urine markers of cardiac risk (i.e., inflammation and oxidative stress).

Eighty adult patients with moderate to severe sleep apnea will be asked to participate. They will have their blood vessel function measured with a non-invasive finger probe, and blood/urine will be collected to measure the cardiac risk markers. Patients will then be 'randomized' to one of two groups: 50% chance that the patient will be asked to take an antioxidant, and a 50% chance that they will be asked to take a placebo tablet (though he/she will not know which one they are taking). After 8 weeks, blood vessel function and markers will be remeasured to determine if antioxidants help patients with sleep apnea.

DETAILED DESCRIPTION:
Purpose: To determine whether treatment of obstructive sleep apnea (OSA) patients with a potent oral antioxidant (alpha lipoic acid, ALA) improves cardiovascular health.

Objectives: The primary objective of the study is to assess the impact of ALA on endothelial function (primary outcome). We will also assess whether ALA improves systemic inflammation and markers of oxidative stress.

Background: Increased production of reactive oxygen species (ROS) and consequent oxidative stress results in tissue damage and activation of inflammation, and is a recognized risk factor for the development of cardiovascular disease (CVD). Obstructive sleep apnea (OSA) is a prevalent under-recognized disorder; moderate to severe disease is found in approximately 9% of randomly selected middle-aged men and 4% of women. In addition, patients with OSA are at increased (i.e., 3 fold) risk of incident CVD including myocardial infarction and acute coronary syndromes. OSA is characterized by repetitive episodes of desaturation followed by reoxygenation; this ischemia/reperfusion is a potent stimulus for the production of ROS, and results in high levels of oxidative stress. Indeed, OSA may be considered a prototypical oxidative stress disease. However, few studies have assessed the potential beneficial impact of antioxidant therapy in OSA patients.

We hypothesize that antioxidants may mitigate some of the adverse CV consequences associated with OSA. The current proposal builds upon our translational work, and focuses on comprehensively assessing the impact of a routinely used potent antioxidant on CV health.

Methods: 80 patients with moderate to severe OSA will be enrolled in a parallel randomized controlled trial (RCT). At baseline, endothelial function will be measured noninvasively using a standard technique (EndoPAT). In addition, we will measure circulating levels of C reactive protein, and markers of oxidative stress (urinary 8-isoprostane and 8-hydroxy-2-deoxy guanosine). Patients will be randomized to either ALA or placebo. Endothelial function and biochemical markers will be remeasured after 12 weeks to determine the impact of ALA.

If ALA does result in significant benefits, this would raise the possibility of using ALA as a therapy in OSA patients to prevent CVD, and justify a larger RCT to validate the result. This is of substantial importance given the high prevalence of OSA in the population.

ELIGIBILITY:
Inclusion Criteria:

* Medically stable adult patients between 35 and 60 years of age with moderate to severe OSA (AHI>15 events/hour by a full night in-laboratory polysomnogram or ambulatory study)
* More than 9 minutes/night spent below oxygen saturation of 90%.
* Subjects who have declined therapy, or who have not adhered to CPAP therapy for at least one month prior to the study recruitment .

Exclusion Criteria:

* Subjects who have excessive daytime sleepiness (Epworth Sleepiness Scale > 12/24)
* Subjects who have documented CVD
* Subjects who have severe sleep associated desaturation (>30% of the sleep study with oxygen saturation <88%).
* Subjects who are on active therapy for OSA or recently treated for OSA with CPAP in the previous month.
* Subjects who have a chronic inflammatory disease (e.g. rheumatoid arthritis, asthma)
* Subjects who regularly use of anti-inflammatory drugs (i.e. systemic or inhaled corticosteroids, statin, ACEI), or other immunosuppressive drugs.
* Subjects who are taking antioxidants.
* Subjects who have diabetes.
* Subjects who have autoimmune syndrome.

Ages: 35 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2022-06-01 (Estimated); Primary Completion 2023-08 (Estimated); Study Completion 2024-08 (Estimated)

PRIMARY OUTCOMES:
Level of C reactive protein (CRP) | 8 weeks
  Level of circulating inflammatory marker
Reactive hyperemia index (RHI) | 8 weeks
  Endothelial function measured by EndoPAT

SECONDARY OUTCOMES:
Plasma level of 8-isoprostane | 8 weeks
  Plasma level of oxidative stress marker of lipid peroxidation
Plasma level of 8-hydroxy-2-deoxy guanosine (8-OHdG) | 8 weeks
  Plasma level of oxidative stress marker of DNA fragmentation
Urinary level of 8-isoprostane | 8 weeks
  Level of oxidative stress marker of lipid peroxidation in urine
Urinary level of 8-hydroxy-2-deoxy guanosine (8-OHdG) | 8 weeks
  Level of oxidative stress marker of DNA fragmentation in urine
Telomere length | 8 weeks
  Telomere length of leukocyte
Augmentation Index (AI) | 8 weeks
  Indirect measure of arterial stiffness measured by EndoPAT

CONTACTS AND LOCATIONS:
Overall Officials: Rachel Jen, MD, Principal Investigator — University of British Columbia
Locations (1):
- UBC Hospital, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No